CLINICAL TRIAL: NCT02792686
Title: ABX464 First in Man, Open Label, Parallel Group, Single Ascending Dose Study
Brief Title: ABX464 First in Man Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX464-001
Record Dates: First submitted 2016-05-30; First posted 2016-06-07 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2016-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — ABX464

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABX464 (Experimental): 50, 100, 150 or 200 mg once a day / Single Administration
  Interventions: Drug: ABX464

INTERVENTIONS:
Drug: ABX464 — Single Administration

SUMMARY:
This study is an open label, parallel group, single ascending dose, exploratory study performed in a single site (Centre Cap, Montpellier, France).

DETAILED DESCRIPTION:
This study is an open label, parallel group, single ascending dose, exploratory study performed in a single site (Centre Cap, Montpellier, France). Six subjects per dose group were enrolled into 1 of 4 groups with escalating doses of ABX464 (50, 100, 150 and 200 mg). For each dose group, a first subject was treated, if no adverse event (AE) occurred, a second subject was dosed one hour later. The four last subjects were dosed the day after if no clinically significant AE occurred. Escalation to the following dose level was decided after review of PK and safety data (laboratory results, ECG, vital signs and AEs)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Subject in good health on the basis of medical history, physical examination, vital signs, electrocardiogram (ECG) and routine laboratory safety tests
* Subject with a BMI of 18 27kg/m²
* Non smokers or light smokers of less than 10 cigarettes per day
* Having given their written informed consent

Exclusion Criteria:

* Subject with any on-going infection or disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients experiencing at least one Adverse Event | Up to 45 days post dosing

SECONDARY OUTCOMES:
Peak Plasma Concentrations (Cmax) of ABX464 and metabolite | Up to 45 days post dosing
Area Under the Curve (AUC) of Plasma Concentrations of ABX464 and metabolite | Up to 45 days post dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Cap, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scherrer D, Rouzier R, Noel Barrett P, Steens JM, Gineste P, Murphy RL, Tazi J, Ehrlich HJ. Pharmacokinetics and tolerability of ABX464, a novel first-in-class compound to treat HIV infection, in healthy HIV-uninfected subjects. J Antimicrob Chemother. 2017 Mar 1;72(3):820-828. doi: 10.1093/jac/dkw458. PMID 27999038